CLINICAL TRIAL: NCT02390843
Title: A Phase 1 Study Using Simvastatin in Combination With Topotecan and Cyclophosphamide in Relapsed and/or Refractory Pediatric Solid and CNS Tumors
Brief Title: Simvastatin With Topotecan and Cyclophosphamide in Relapsed and/or Refractory Pediatric Solid and CNS Tumors
Acronym: AflacST1402
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Children's Healthcare of Atlanta (Other)
Responsible Party: Principal Investigator, Kelly Goldsmith, Assistant Professor, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00078790
Record Dates: First submitted 2015-02-24; First posted 2015-03-18 (Estimated); Last update posted 2020-04-03 (Actual); Status verified 2020-04

CONDITIONS: Retinoblastoma; Clear Cell Sarcoma; Renal Cell Carcinoma; Rhabdoid Tumor; Wilms Tumor; Hepatoblastoma; Neuroblastoma; Germ Cell Tumors; Ewings Sarcoma; Non-rhabdomyosarcoma Soft Tissue Sarcoma; Osteosarcoma; Rhabdomyosarcoma
MeSH Terms: conditions — Retinoblastoma; Sarcoma, Clear Cell; Carcinoma, Renal Cell; Rhabdoid Tumor; Wilms Tumor; Hepatoblastoma; Neuroblastoma; Neoplasms, Germ Cell and Embryonal; Sarcoma, Ewing; Sarcoma; Osteosarcoma; Rhabdomyosarcoma | interventions — Simvastatin; Cyclophosphamide; Topotecan; Granulocyte Colony-Stimulating Factor; pegylated granulocyte colony-stimulating factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- simvastatin + topotecan/cyclophosphamide (Experimental): During dose escalation (phase I), standard 3+3 design will be followed.
  Interventions: Drug: Simvastatin; Drug: Cyclophosphamide; Drug: Topotecan; Drug: Myeloid growth factor

INTERVENTIONS:
Drug: Simvastatin — The starting dose of simvastatin will be 140 mg/m^2/dose BID for 21 days for the first group. Dose escalation for subsequent groups will be 180 mg/m^2/dose BID, 225 mg/m^2/dose BID, and 290 mg/m^2/dose BID. If the maximum tolerated dose (MTD) has been exceeded at the first dose level, then the subsequent cohort of subjects will be treated at a dose of 100 mg/m2/dose BID (dose level 0). Simvastatin will be administered orally twice daily, approximately 12 hours apart. Feeding tube (nasogastric tube or gastrostomy tube, NOT a jejunum localized tube) administration is allowed. If a subject vomits a dose of simvastatin, it will not be repeated.
  Other Names: zocor
Drug: Cyclophosphamide — The dose of cyclophosphamide will be fixed at 250 mg/m^2/dose. Cyclophosphamide will be administered intravenously over 30 minutes once daily for 5 days every 21 days.
  Other Names: Cytoxan; Neosar
Drug: Topotecan — The dose of topotecan will be fixed at 0.75 mg/m^2/dose. Topotecan will be administered, after cyclophosphamide, intravenously over 30 minutes once daily for 5 days every 21 days.
  Other Names: Hycamtin
Drug: Myeloid growth factor — Myeloid growth factor (G-CSF or pegylated G-CSF) will be initiated 24-48 hours after the completion of topotecan and cyclophosphamide for all subjects, which would be day 6 or 7. Myeloid growth factor should continue until the absolute neutrophil count is greater than 2,000/mm^3
  Other Names: Granulocyte colony-stimulating factor (G-CSF); pegylated granulocyte colony-stimulating factor

SUMMARY:
This is a Phase I trial with new experimental drugs such as simvastatin in combination with topotecan and cyclophosphamide in the hopes of finding a drug that may work against tumors that have come back or that have not responded to standard therapy. This study will define toxicity of high dose simvastatin in combination with topotecan and cyclophosphamide and evaluate for cholesterol levels and IL6/STAT3 pathway changes as biomarkers of patient response.

DETAILED DESCRIPTION:
Chemotherapy resistance is a major cause of treatment failure in pediatric solid tumors. STAT3 (Signal Transducer and Activator of Transcription 3) is a transcription factor that promotes tumor proliferation, metastasis and chemotherapy resistance. Pediatric solid tumors such as neuroblastoma, rhabdomyosarcoma, osteosarcoma, Ewing sarcoma, and central nervous system (CNS) tumors such as glioblastoma and medulloblastoma have aberrant STAT3 signaling. In neuroblastoma, bone marrow production of interleukin 6 (IL-6), a STAT3 activating cytokine, is associated with poor prognosis. Thus STAT3 and its cognate ligand, IL-6, are rational therapeutic targets in pediatric solid and CNS tumors. HMG-CoA (3-hydroxy-3-methylglutaryl-coenzyme A) reductase inhibitors, or "statins", lower LDL (low density lipoprotein) cholesterol by inhibiting the rate-limiting step in cholesterol biosynthesis. Pleiotropic properties of statins have been found to not only contribute to lowering the risk of heart disease, but decrease the incidence of cancer as well, leading to their use in clinical trials for adult solid and CNS tumors. Statins have been shown to inhibit IL-6 mediated STAT3 activation to prevent the recruitment of pro-inflammatory cells to injured heart tissue in adult patients. Therefore, the investigators hypothesize that the HMG-CoA reductase inhibitor, simvastatin, will augment chemotherapy effects to improve survival of patients with refractory or relapsed pediatric solid and CNS tumors. This is a Phase I trial of simvastatin in combination with topotecan and cyclophosphamide for refractory and/or relapsed solid or CNS tumors of childhood, in which the investigators will define toxicity and evaluate cholesterol levels and IL6/STAT3 pathway changes as biomarkers of patient response.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have had histologic verification of malignancy at original diagnosis or relapse. All subjects with relapsed or refractory solid tumors are eligible including primary or metastatic CNS tumors. In the case of diffuse intrinsic pontine glioma (DIPG), or optic pathway glioma, imaging findings consistent with these tumors will suffice without the need for biopsy for histologic verification.
* Subjects must have either measurable (the presence of at least one lesion that can be accurately measured in at least one dimension with the longest diameter at least 20 mm. With spiral CT scan, lesions must be at least 10 mm.) or evaluable disease (the presence of at least one lesion that cannot be accurately measured in at least one dimension. Such lesions may be evaluable by nuclear medicine techniques, immunocytochemistry techniques, tumor markers or other reliable measures.)
* Subject's current disease state must be one for which there is no known curative therapy.
* Karnofsky ≥ 60% for subjects > 16 years of age and Lansky ≥ 50 for subjects ≤ 16 years of age
* Subjects must have fully recovered from the acute toxic effects of all prior anti-cancer chemotherapy

  1. Myelosuppressive chemotherapy: At least 21 days after the last dose of myelosuppressive chemotherapy (42 days if prior nitrosourea).
  2. Hematopoietic growth factors: At least 14 days after the last dose of a long-acting growth factor (e.g. Pegfilgrastim) or 7 days for short acting growth factor. For agents that have known adverse events occurring beyond 7 days after administration, this period must be extended beyond the time during which adverse events are known to occur. The duration of this interval must be discussed with the study chair.
  3. Biologic (anti-neoplastic agent): At least 7 days after the last dose of a biologic agent. For agents that have known adverse events occurring beyond 7 days after administration, this period must be extended beyond the time during which adverse events are known to occur. The duration of this interval must be discussed with the study chair.
  4. Immunotherapy: At least 42 days after the completion of any type of immunotherapy, e.g. tumor vaccines.
  5. Monoclonal antibodies: At least 3 half-lives of the antibody after the last dose of a monoclonal antibody.
  6. external beam radiation therapy (XRT): At least 14 days after local palliative XRT (small port); 6 weeks must have elapsed since treatment with therapeutic doses of I131-meta-iodobenzylguanidine (MIBG); At least 150 days must have elapsed if prior total body irradiation (TBI), craniospinal XRT, or if ≥ 50% radiation of pelvis; At least 42 days must have elapsed if other substantial bone marrow (BM) radiation.
  7. Stem Cell Infusion without TBI: No evidence of active graft vs. host disease and at least 84 days must have elapsed after transplant and 42 days for autologous stem cell infusion after I131-MIBG therapy.
  8. Subjects must not have received any prior therapy with simvastatin.
* Adequate Bone Marrow Function Defined as:

  1. For subjects with solid tumors without known bone marrow involvement: Peripheral absolute neutrophil count (ANC) ≥ 750/mm3, Platelet count ≥ 75,000/mm3 (transfusion independent, defined as not receiving platelet transfusions for at least 7 days prior to enrollment)
  2. Subjects with known bone marrow metastatic disease will be eligible for study provided they meet the blood counts in a. (may receive transfusions provided they are not known to be refractory to red cell or platelet transfusions). These subjects will not be evaluable for hematologic toxicity. If dose-limiting hematologic toxicity is observed, all subsequent subjects enrolled must be evaluable for hematologic toxicity.
* Adequate Renal Function Defined as:

  1. Creatinine clearance or radioisotope glomerular filtration rate (GFR) 70ml/min/1.73 m^2 or
  2. A serum creatinine based on age/gender as follows:
* Age: 1 to < 2 years; Male and female serum creatinine: 0.6 mg/dL
* 2 to < 6 years; Male and female serum creatinine: 0.8 mg/dL
* 6 to < 10 years; Male and female serum creatinine: 1.0 mg/dL
* 10 to < 13 years; Male and female serum creatinine: 1.2 mg/dL
* 13 to < 16 years; Male serum creatinine: 1.5 mg/dL and female serum creatinine: 1.4 mg/dL
* ≥ 16 years; Male serum creatinine: 1.7 mg/dL and female serum creatinine: 1.4 mg/dL
* Adequate Liver Function Defined as:

  1. Bilirubin (sum of conjugated + unconjugated) ≤ 1.5 x upper limit of normal (ULN) for age
  2. serum glutamate pyruvate transaminase (SGPT) or ALT ≤ 135 U/L. For the purpose of this study, the ULN for SGPT is 45 U/L.
* Adequate Cardiac Function Defined as: corrected QT interval (QTc) ≤ 480 msec
* Normal Creatinine Phosphokinase (CPK) Defined As Not Exceeding Maximum Value:
* Age: 0 to < 4 years; Male and female maximum CPK : 305 units/L
* 4 to < 7 years; Male and female maximum CPK : 230 units/L
* 7 to < 10 years; Male and female maximum CPK : 365 units/L
* 10 to < 12 years; Male maximum CPK: 215 units/L and female maximum CPK: 230 units/L
* 12 to < 14 years; Male maximum CPK: 330 units/L and female maximum CPK: 295 units/L
* 14 to < 16 years; Male maximum CPK: 335 units/L and female maximum CPK: 240 units/L
* 16 to < 19 years; Male maximum CPK: 370 units/L and female maximum CPK: 230 units/L
* ≥ 19 years; Male maximum CPK: 170 units/L and female maximum CPK: 145 units/L
* Willing to sign consent or assent/primary caregiver willing to give consent

Exclusion Criteria:

* Pregnancy or breast-feeding
* Concomitant medication dependency including corticosteroids, investigational drugs, anti-cancer agents, anti-graft-versus-host disease (GVHD) agents post-transplant
* subjects who are unable to swallow a tablet or liquid must have a nasogastric (NG) or gastric (G) tube through which the medicine can be administered
* subjects receiving known cytochrome P450 3A4 (CYP3A4) Inhibitors or Inducers
* subjects with uncontrolled infection
* subjects who received prior solid organ transplantation
* subjects with current or previous treatment with 3-hydroxy-3-methylglutaryl-coenzyme A (HMG CoA) reductase inhibitor (any statin)

Ages: 1 Year to 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 13 (Actual)
Dates: Start 2015-02; Primary Completion 2019-09-22 (Actual); Study Completion 2019-09-22 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of Simvastatin | First treatment to toxicity (up to 24 months)
  MTD will be the maximum dose at which fewer than one-third of subjects experience dose-limiting toxicities (DLTs) during Cycle 1 of therapy.
Number of Dose-Limiting Toxicities (DLTs) | Up to 24 months
  DLT will be defined as any of the following events that are possibly, probably, or definitely attributable to study drug:
  Non-hematological dose-limiting toxicity: Any Grade 3 or 4 non-hematological toxicity (excluding nausea, alanine transaminase (ALT) or aspartate aminotransferase (AST) that returns to baseline or ≤ grade 1 within 7 days of study drug interruption, fever, infection, hypophosphatemia, hypokalemia, hypocalcemia, hypomagnesemia, or creatinine phosphokinase (CPK) elevation that returns to baseline or ≤ grade 1 within 7 days of study drug interruption), Any Grade 2 non-hematological toxicity that persists for ≥ 7 days and is considered sufficiently medically significant or sufficiently intolerable by subjects that it requires treatment interruption, or hematological dose-limiting toxicity, defined as neutropenia or thrombocytopenia that precludes initiation of the next cycle of therapy within 14 days of the scheduled start date.

SECONDARY OUTCOMES:
Percentage of Participants With Overall Tumor Response (Response Rate) | 24 months
  Response is defined as CR (Complete Response) or PR (Partial Response) per Response Evaluation Criteria in Solid Tumor (RECIST criteria). Possible evaluations include: CR: Disappearance of all target lesions. PR: At least a 30% decrease in the size of target lesions.
  Response rate (%) = (number of patients with CR+PR/number of patients)*100
Change in Total Cholesterol Level | Baseline, 24 months
  Change in serum total cholesterol level after treatment with simvastatin. A decrease from baseline to the end of treatment, a negative value, indicates an improvement.
Change in serum interleukin-6 (IL-6) level | Baseline, 24 months
  Change in serum interleukin-6 (IL-6) level after treatment with simvastatin. Serum levels of the IL-6 will be assayed using by enzyme-linked immunosorbent assay (ELISA). Higher levels are typically interpreted as worsening of condition.
Change in soluble interleukin 6 receptor (sIL-6R) | Baseline, 24 months
  Change in serum interleukin-6 (IL-6) level after treatment with simvastatin. Serum levels of the sIL-6r will be assayed using by enzyme-linked immunosorbent assay (ELISA). Higher levels are typically interpreted as worsening of condition.
Change in signal transducer and activator of transcription 3 (STAT-3) expression | Baseline, 24 months
  Change in STAT-3 expression after treatment with simvastatin. STAT-3 will be measured using phospho-specific flow cytometry, or phospho-flow.
Change in phospho-STAT3 expression | Baseline, 24 months
  Change in phospho-STAT3 expression after treatment with simvastatin. Phospho-STAT3 expression will be measured using phospho-specific flow cytometry, or phospho-flow.

CONTACTS AND LOCATIONS:
Overall Officials: Kelly Goldsmith, MD, Principal Investigator — Emory University/Children's Healthcare of Atlanta
Locations (1):
- Children's Healthcare of Atlanta/Emory University, Atlanta, Georgia, United States

REFERENCES:
- [Derived] Hattinger CM, Patrizio MP, Magagnoli F, Luppi S, Serra M. An update on emerging drugs in osteosarcoma: towards tailored therapies? Expert Opin Emerg Drugs. 2019 Sep;24(3):153-171. doi: 10.1080/14728214.2019.1654455. Epub 2019 Aug 14. PMID 31401903